CLINICAL TRIAL: NCT03358056
Title: Effects of Mindfulness Based Cognitive Therapy on Emotional Processing
Acronym: MESI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/7185/I
Record Dates: First submitted 2017-10-17; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Unipolar Depression; Anxiety Disorders; Adjustment Disorders; Emotional Instability
Keywords: Mindfulness; Emotion; Mindfulenss-based cognitive therapy
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Adjustment Disorders | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-based Cognitive Therapy (Experimental)
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — Mindfulness-based cognitive therapy (MBCT) is a manualized, 8 weeks-group-based training derived from mindfulness-based stress reduction (MBSR) and cognitive-behavioral therapy (CBT). In MBCT participants are trained in how to be more aware of their bodily sensations, thoughts and feelings associated with negative emotional states. Mindfulness exercises and cognitive-behavioral skills are practiced both during the sessions and through homework assignments. The program is structured in 2.30 h group sessions over 8 consecutive weeks.

SUMMARY:
Background: In the last 30 years mindfulness-based approaches have been extensively used for a variety of mental disorders, including affective disorders characterized by emotional instability. Mindfulness based cognitive therapy (MBCT) is an 8-week intervention that combines mindfulness practices with cognitive behavioural therapy. Although changes in emotional processing have been postulated as one of mindfulness mechanisms of action, the effects of mindfulness-based programs on objective tasks of emotional processing have been poorly studied.

Objective: To explore the effects of mindfulness-based cognitive therapy (MBCT) on emotional processing in a sample of individuals with emotional instability attended in a mental-health public service.

Methods: The sample (n = 30) will be recruited from public mental-health outpatient centers in Barcelona, Spain. Inclusion criteria: 1) high emotional instability defined as scores above 96 on the Difficulties in Emotion Regulation Scale (DERS), 2) age between 18 and 65 years, 4) no prior experience with mindfulness/meditation. Exclusion criteria: 1) risk of suicide (attempted suicide in the last year or current suicidal ideation). Psychotropic medication will be permitted, as long as there are no changes in dose/type during the study period.

Measures Diagnostic measures (MINI, DERS, CGI) and a complete medical register will be collected prior inclusion in the study. Additional measures on personality (ZKPQ) and temperament (Temps-A) will be collected as well.

Primary outcome:

Emotional processing task: Participants will complete the FERT task at two time points: baseline (pre-treatment) and 8 weeks (post-treatment).

Secondary outcomes:

In addition, participants will complete the following assessments (pre-and-post- treatment):

* Depressive Symptoms (QIDS-16)
* Anxiety Symptoms (STAI)
* Mindfulness (FFMQ and EQ).

Treatment Mindfulness-based cognitive therapy (MBCT) is a manualized, 8 weeks-group-based training derived from mindfulness-based stress reduction (MBSR) and cognitive-behavioral therapy (CBT). In MBCT participants are trained in how to be more aware of their bodily sensations, thoughts and feelings associated with negative emotional states. Mindfulness exercises and cognitive-behavioral skills are practiced both during the sessions and through homework assignments. The program is structured in 2.30 h group sessions over 8 consecutive weeks.

DETAILED DESCRIPTION:
BACKGROUND

Mindfulness is typically defined as a present-centered non-judgmental awareness (Kabat-Zinn, 1990). In the last 30 years mindfulness-based approaches have been extensively used for a variety of mental disorders, including affective disorders characterized by emotion dysregulation (Khoury et al., 2013).

Mindfulness-based cognitive therapy (MBCT) includes meditation techniques to help participants become more aware of their experience in the present moment. Participants learn the practice of mindfulness meditation through 8 classes held on a weekly basis. Unlike other mindfulness-based approaches, MBCT also includes basic exercises derived from cognitive therapy that demonstrate the links between thinking and feeling and how participants can care for themselves (Williams & Kuyken, 2012). Although the efficacy of MBCT has been established in a number of studies (Barnhofer et al., 2009; Kuyken et al., 2008; Ma & Teasdale, 2004), little is known in regard to the mechanisms underlying mindfulness beneficial effects. Holzel (Holzel et al., 2011) suggests that one of these mechanisms is related to the effects of mindfulness in emotion regulation, however this mechanism has been poorly studied, especially in clinical samples. Therefore the aim of the present study is to explore the performance of a naturalistically recruited sample of patients with high emotional instability in a task of facial expression recognition. We hypothesized that mindfulness practice will lead to changes in emotional processing as measured with the facial emotion recognition task (FERT).

OBJECTIVES Primary aim: The objective of the present study is to investigate the effects of MBCT on emotional processing in a sample of individuals with emotion instability attended in a mental-health public service.

Secondarily, the effect of MBCT on depressive and anxiety symptoms and mindfulness capacities will be assessed.

METHOD:

This is a pre-post interventional study. Given the exploratory nature of this study a sample of 30 participants will be recruited from public mental-health outpatient centers in Barcelona, Spain located at the catchment area of the PSMAR (CSMA Sant Martí Sud, CSMA Sant Martí Nord, CSMA Santa Coloma y CSMA La Mina). Inclusion criteria: 1) high emotional instability defined as scores above 76 on the Difficulties in Emotion Regulation Scale (DERS), 2) age between 18 and 65 years, 3) no prior experience with mindfulness/meditation. Exclusion criteria: 1) risk of suicide (attempted suicide in the last year). Psychotropic medication will be permitted, as long as there are no changes in dose/type during the study period.

• Measures

Diagnostic measures:

Psychiatric symptoms will be collected with the Psychiatric Diagnostic Screening Questionnaire (PDSQ; Pérez Gálvez, García Fernández, de Vicente Manzaro, & Olivera Valenzuela, 2010; Zimmerman & Mattia, 2001) in order to obtain Axis I comorbidities. The PDSQ contains 13 sub-scales screening for: major depressive disorder, bulimia, post-traumatic stress disorder, panic disorder, agoraphobia, social phobia, generalized anxiety disorder, obsessive-compulsive disorder, alcohol abuse/dependence, drug abuse/dependence, somatization, hypochondriasis and psychosis. A complete medical register will be also collected prior inclusion in the study.

The Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004; Hervás & Jódar, 2008) will be used for assessing emotional instability. Participants will be included in the study if they scored higher than 76 (1 SD above the mean of the general population). The DERS is a 28 item-questionnaire that provides a total score and 4 sub-scores measuring: non-acceptance of emotional responses, lack of emotional awareness, lack of emotional clarity and limited access to emotion regulation strategies.

Clinical Global Impression Severity and Improvement (CGI-S and CGI-I; Kadouri, Corruble, & Falissard, 2007). The CGI-S scale would be used to evaluate the clinical severity of the participant in a scale from 1 to 7 ("not ill at all", to "very ill"). The CGI will be clinician-administered and self-reported. In addition, the CGI-I will be also used, in order to evaluate the improvement between the baseline visit and the post-intervention assessment (from 1: "very slight deterioration" to 7: "maximum deterioration").

The TEMPS-A scale (Vázquez and Akiskal 2005) is a self-evaluation questionnaire used to assess the four basic affective temperaments (hyperthymic, depressive, cyclothymic, and irritable), and the anxious temperament.

Primary outcome:

Emotional processing task: Participants will complete the Facial Expression Recognition Task (FERT) task at two time points: baseline (pre-treatment) and 8 weeks (post-treatment). The FERT uses stimuli pictures of faces expressing basic emotions (i.e., anger, disgust, fear, happiness, sadness and surprise) from 10 actors. Each emotion was morphed, in 10% steps, between two standard images of 0% (neutral) and 100 % (full emotion). Four examples of each emotion at each intensity (10-100%) are presented (6 emotions x 10 intensities x 4 actor examples = 240 stimuli). Each face is also presented in a neutral expression, so there are a total of 250 stimulus presentations. Facial expressions appear on the screen for 500ms, followed by a blank screen. Participants are asked to classify the expression of presented faces as quickly and accurately as possible by clicking in one of the seven labeled emotion keys. The next face is not presented until an expression has been assigned to the previous face. Accuracy and reaction time are recorded.

Secondary outcomes:

In addition, participants will complete the following questionnaires (pre-and-post- treatment):

Depressive Symptoms (QIDS-16; Rush et al., 2003). Self-reported 16 item questionnaire that assess depressive symptoms.

Anxiety Symptoms (STAI; Spielberg, 1983). To assess anxiety symptoms the state version of the STAI will be used.

Mindfulness (FFMQ and EQ). The Five Facet Mindfulness Questionnaire (Baer, Smith, Hopkins, Krietemeyer, & Toney, 2006; Cebolla et al., 2012). The FFMQ measures five different factors: (1) Observe, (2) Describe, (3) Acting with awareness, (4) Non-judging the inner experience and (5) Non-reacting to the inner experience. Participants were asked to rate the degree of concordance with each statement on a 5-point Likert scale that ranges from 1 (never or very rarely, true) to 5 (very often or always, true). The Experiences Questionnaire (Fresco et al., 2007; Soler et al., 2014). This instrument comprises 11 items and measures decentering, defined as the capacity to observe one's thoughts and emotions as temporary events of the mind. The EQ items are scored in a 5-point-Likert-type scale, ranging from never to all the time, with higher scores indicating more decentering.

* Treatment Mindfulness-based cognitive therapy (MBCT; Segal, Williams, & Teasdale, 2002)) is a manualized, 8 weeks-group-based training derived from mindfulness-based stress reduction (MBSR) and cognitive-behavioral therapy (CBT). In MBCT participants are trained in how to be more aware of their bodily sensations, thoughts and feelings associated with negative emotional states. Mindfulness exercises and cognitive-behavioral skills are practiced both during the sessions and through homework assignments. The program is structured in 2.30 h group sessions over 8 consecutive weeks.
* Procedure. Participants who fulfil inclusion/exclusion criteria will be invited to participate in the study. After explaining study's procedures, participants will receive the "Participant Information Sheet" and the informed consent will be signed. Thereafter, participants will complete the FERT task using a tablet and paper-and-pencil questionnaires. Baseline assessments will be conducted within one week prior to the start of the group-therapy. Assessments (FERT task and questionnaires) will be completed at post-treatment, also within a week of concluding the group. A detailed description of the measures used by study phase can be found in Table 1.

ELIGIBILITY:
Inclusion Criteria:

* high emotional instability defined as scores above 96 on the Difficulties in Emotion Regulation Scale (DERS)
* diagnosis of unipolar affective disorders
* age between 18 and 65 years
* no prior experience with mindfulness/meditation

Exclusion Criteria:

* risk of suicide (attempted suicide in the last year or current suicidal ideation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Facial Emotion Recognition Task | 8 past weeks
  Computarized facial emotion recognition task

SECONDARY OUTCOMES:
Quick Depression Inventory | 1 past week
  Inventory for assessing depressive symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Parc de Salut Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided